CLINICAL TRIAL: NCT04111640
Title: Evaluation of the Effectiveness of a Computerized Cognitive Training in the Early Stages of Neurodegenerative Diseases
Brief Title: Computerized Cognitive Training in Neurodegenerative Diseases (NDD2019)
Acronym: NDD2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NDD2019
Record Dates: First submitted 2019-09-12; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Mild Cognitive Impairment
Keywords: neurodegenerative diseas; non-pharmacological treatments; cognitive training
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel assignment, prospective, double-blind, randomized, controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A computer-supported cognitive training for the training of logical-executive and working-memory functions (CoRe software)
  Interventions: Other: Control Group
- Control Group (Other): Paper and pencil cognitive training (paper-and-pencil CoRe version)
  Interventions: Other: CoRe software

INTERVENTIONS:
Other: CoRe software — Computer-supported cognitive training (CT)
  Arms: Control Group
Other: Control Group — Paper and pencil cognitive training (paper-and-pencil CoRe version)
  Arms: Experimental group

SUMMARY:
The prevalence of neurodegenerative diseases is expected to increase over the next years, in parallel to the aging of the world population. Therefore, research efforts need to be devoted to evaluate intervention strategies that delay the onset of cognitive decline. Given the paucity of pharmacological interventions, strategies for non-pharmacological enhancement, such as cognitive training, are receiving increasing attention. Moreover, the advances in the development of Information & Communication Technologies (ICT) has recently prompted the possibility to develop computer-based solution, also called Serious Game (SG), for the training of one or more cognitive functions. This approach could help overcome the limits of traditional paper-and-pencil cognitive intervention techniques. However, the clinical, ethical, economic and research impact of the use of these computer-based solutions in these target populations is still under discussion. In order to acquire more academic and professional credibility and acceptance, researchers need to collect more data to test and evolve usability and usefulness of SG as clinical tools targeting people with dementia-related disorders.

The general aim of this research is to evaluate the effects of a computer-supported Cognitive Training (CT) compared to a paper-and-pencil CT, in the early stage of neurodegenerative diseases. Patients with Mild Cognitive Impairment (MCI) are enrolled and randomly assigned to the experimental group (CoRe software) or control group (paper-and-pencil CoRe version). All patients are evaluated before (T0) and after (T1) treatment with an exhaustive neuropsychological assessment. Furthermore, follow-up visits are scheduled 6 months (T2) and 12 months (T3) after the end of the treatment.

DETAILED DESCRIPTION:
Serious games (SG), are digital applications specialized for purpose other than entertaining. These technology devices could help to overcome the limits of traditional paper-and-pencil approaches. These traditional interventions, even if particular familiar to older patients, involve indeed some disadvantages, such as data management and analysis particularly complex for therapists; possible learning effects related to stimuli, boredom and reduction of the patient's compliance.

Conversely, SG uses motivational cues and provides real-time feedback; task complexity and response time demands may change frequently during and across sessions, in accordance with changes in individual performance. This allows to avoid over- or under-stimulation and to train areas of relative weakness. Computer support also saves time for therapists in the preparation of exercises and allows to record all session parameters for further statistics. Talking about disadvantages, the more critical is that elderly people might have poor information technology skills with a consequent lack of familiarity with technological devices. These difficulties derive from the fact that most of the SG used have been developed for entertainment purposes (e.g., the Nintendo Wii Fit, Wii Sports, and Big Brain Academy) and for a "typical healthy user" in mind. Some practical recommendations for the usability and usefulness of SG as clinical tools in dementia-related disorders were collected, but there is still no a general consensus about how, when and for what purpose these digital games should be developed. In fact, in the contest of neurodegenerative disease, cognitive intervention to be effective must be proportionate to the degree of cognitive deterioration and consequently it is necessary to take into account the phases of the disease, the speciﬁc disease characteristics and the speciﬁc cognitive domains affected. Some studies suggested that computerized CT is efficacious at the early phases of the disease, or where MCI is present, while it may not be beneficial at the dementia stage. Though these emerging results are encouraging, some issue about the use of this computer-based solution as clinical tools remain unresolved.

In this frame, we develop a computer-based CT (CoRe software) for the training of logical-executive and working-memory functions. We aim to assess the efficacy of this computer-supported CT compared to a paper-and-pencil CoRe version. This could be useful for two main reasons: 1) understand the comparability of the two interventions; 2) explore possible extra advantages of the CoRe software with respect to the paper-and-pencil version that could make it more suitable for the clinical routine.

CoRe is an ontology-based software tool that allows several degrees of personalization and the possibility to generate different patient-tailored exercises; for a more detailed description see previous papers.

Inpatients with idiopathic PD are recruited from the Neurorehabilitation Unit of the IRCCS Mondino Foundation. The diagnosis of mild dementia or PD-MCI is formulated on the basis of a comprehensive neuropsychological evaluation (baseline cognitive assessment - T0) according to the guidelines presented in the literature. The following standardized tests assessing different domains are used:

* global cognitive function: Mini-Mental State Examination (MMSE) and Montreal Montreal Overall Cognitive Assessment (MoCA);
* memory: verbal (Verbal Span; Digit Span) and spatial (Corsi's blocktapping test - CBTT) span; verbal long-term memory (Logical Memory Test immediate and delayed recall; Rey's 15-word test immediate and delayed recall); spatial long-term memory (Rey Complex Figure delayed recall - RCF-dr);
* logical-executive functions: non-verbal reasoning; frontal functionality (Frontal Assessment Battery - FAB); semantic fluency (animals, fruits, car brands), phonological fluency (FAS);
* attention: visual selective attention (Attentive Matrices); simple speed processing and complex attention (Trail Making Test parts A - TMT A and part B - TMT B);
* visuospatial abilities: constructive apraxia Rey Complex Figure copy - RCF-copy.

The same battery is also used at the post-training assessment (T1) and at the follow-up visits six months (T2) and one year after (T3). Parallel versions are applied when available (verbal long-term memory tests), in order to avoid the learning effect. All the test scores are corrected for age, sex, and education and compared with the values available for the Italian population.

At the baseline, the cognitive reserve is assessed using Cognitive Reserve Index questionnaire (CRIq). The patients' functional status is assessed using Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) at the baseline and at the last follow-up visit after one year (T3). Moreover, mood is assessed using the Beck Depression Inventory (BDI) at the baseline and at the follow-up visits (T1, T2 and T3), while quality of life is assessed using the 36-Item Short Form Health Survey questionnaire (SF-36) at the baseline and at the follow-up visits six months (T2) and one year (T3) after training.

This study is a prospective, double-blind Randomized Controlled Trial. All the patients recruited undergo baseline cognitive assessment (T0). Patients who meet the inclusion and exclusion criteria are enrolled and randomly assigned to the experimental group (CoRe software) or control group (paper-and-pencil CoRe version). CT program consists of 12 individual sessions (3 sessions/week) each lasting 45 minutes of computer-based or paper-and-pencil logical-executive and working-memory tasks.

All the patients are evaluated at the end of the 3-weeks training (T1), to detect the training effect, and six month (T2) and one year (T3) after the end of CT to assess the persistence of the training-related improvement and also to evaluate the impact of CT on the evolution of cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD according to UKPDBB criteria (Hughes, Daniel, Kilford, & Lees, 1992) and Hoehn&Yahr scale≤4 (Hoehn & Yahr, 1967);
* presence of PD-MCI single-domain (executive) or PD-MCI multiple-domain with executive involvement (Litvan et al., 2012);
* age between 50 and 85 years;
* education level ≥5 years.

Exclusion Criteria:

* pre-existing cognitive impairment (e.g. aphasia,neglect);
* severe disturbances in consciousness;
* severe sensory or motor disturbances that do not allow the patient to control the trunk or to maintain the sitting position; in particular patients with disturbing resting and/or action tremor (corresponding to score 2-4 in the specific items of Unified Parkinson's Disease Rating Scale (UPDRS III) (Fahn,1987) were excluded;
* concomitant severe psychiatric or neurological conditions;
* patients with Deep Brain Stimulation.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Global cognitive functioning measured by Mini-Mental State Examination (MMSE) | After 3 -week rehabilitative program (T1), 6 months (T2) and 1 year (T3) after the end of rehabilitation program
  It is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. The score is between 0-30. Lower score is worse cognitive functioning.
Change in Global cognitive functioning measured by Montreal Overall Cognitive Assessment (MoCA) | After 3 -week rehabilitative program (T1), 6 months (T2) and 1 year (T3) after the end of rehabilitation program
  It is a widely used screening assessment for detecting cognitive impairment. It assesses several cognitive domains:
  The short-term memory recall task (5 points). Visuospatial abilities a clock-drawing task (3 points) and a three-dimensional cube copy (1 point).
  Multiple aspects of executive functions are assessed using an alternation task adapted from the trail-making B task (1 point), a phonemic fluency task (1 point), and a two-item verbal abstraction task (2 points).
  Attention, concentration, and working memory are evaluated using a sustained attention task ( 1 point), a serial subtraction task (3 points), and digits forward and backward (1 point each).
  Language is assessed using a three-item confrontation naming task with low-familiarity animals (3 points), repetition of two syntactically complex sentences (2 points), and the aforementioned fluency task.
  Finally, orientation to time and place (6 points). Low score is worse outcome.

SECONDARY OUTCOMES:
Change in Memory | after 3 -week rehabilitative program (T1), 6 months (T2) and 1 year (T3) after the end of rehabilitation program
  Verbal and spatial span; verbal long-term memory; spatial long-term memory by using scales. Higher scores are better outcomes
Change in executive functions | after 3 -week rehabilitative program (T1), 6 months (T2) and 1 year (T3) after the end of rehabilitation program
  Logical-executive functions; attention; visuospatial abilities by using scales. Higher scores are better outcomes
Change in Mood (assessed by Beck Depression Inventory - BDI) | after 3 -week rehabilitative program (T1), 6 months (T2) and 1 year (T3) after the end of rehabilitation program
  Contains 21 questions. The items are rated on a 4-point severity scale (0-3) and are summed to give a total score (range 0-63). A higher score denotes more severe depression.
Change in Quality of life (assessed by Short Form-36 Health Survey - SF-36) | after 3 -week rehabilitative program (T1), 6 months (T2) and 1 year (T3) after the end of rehabilitation program
  Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Low score is worse quality of life.
Change in The evolution of cognitive profile (assessed by Clinical Dementia Rating Scale - CDR) | after 3 -week rehabilitative program (T1), 6 months (T2) and 1 year (T3) after the end of rehabilitation program
  CDR is a widely utilized clinical tool for grading the relative severity of dementia with scores that range from 0 (no impairment) to 3 (severe impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sinforiani, MD, Principal Investigator — IRCCS Mondino Foundation, Pavia
Locations (1):
- Struttura Semplice Neuropsicologia Clinica/ Centro UVA, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayeux R, Stern Y. Epidemiology of Alzheimer disease. Cold Spring Harb Perspect Med. 2012 Aug 1;2(8):a006239. doi: 10.1101/cshperspect.a006239. PMID 22908189
- [Background] Belleville S. Cognitive training for persons with mild cognitive impairment. Int Psychogeriatr. 2008 Feb;20(1):57-66. doi: 10.1017/S104161020700631X. Epub 2007 Oct 25. PMID 17958927
- [Background] Jean L, Bergeron ME, Thivierge S, Simard M. Cognitive intervention programs for individuals with mild cognitive impairment: systematic review of the literature. Am J Geriatr Psychiatry. 2010 Apr;18(4):281-96. doi: 10.1097/JGP.0b013e3181c37ce9. PMID 20220584
- [Background] Robert PH, Konig A, Amieva H, Andrieu S, Bremond F, Bullock R, Ceccaldi M, Dubois B, Gauthier S, Kenigsberg PA, Nave S, Orgogozo JM, Piano J, Benoit M, Touchon J, Vellas B, Yesavage J, Manera V. Recommendations for the use of Serious Games in people with Alzheimer's Disease, related disorders and frailty. Front Aging Neurosci. 2014 Mar 24;6:54. doi: 10.3389/fnagi.2014.00054. eCollection 2014. PMID 24715864
- [Background] Walton CC, Naismith SL, Lampit A, Mowszowski L, Lewis SJ. Cognitive Training in Parkinson's Disease. Neurorehabil Neural Repair. 2017 Mar;31(3):207-216. doi: 10.1177/1545968316680489. Epub 2016 Dec 13. PMID 27899737
- [Background] Coyle H, Traynor V, Solowij N. Computerized and virtual reality cognitive training for individuals at high risk of cognitive decline: systematic review of the literature. Am J Geriatr Psychiatry. 2015 Apr;23(4):335-359. doi: 10.1016/j.jagp.2014.04.009. Epub 2014 May 14. PMID 24998488
- [Background] Bernini S, Alloni A, Panzarasa S, Picascia M, Quaglini S, Tassorelli C, Sinforiani E. A computer-based cognitive training in Mild Cognitive Impairment in Parkinson's Disease. NeuroRehabilitation. 2019;44(4):555-567. doi: 10.3233/NRE-192714. PMID 31256092
- [Background] Alloni A, Quaglini S, Panzarasa S, Sinforiani E, Bernini S. Evaluation of an ontology-based system for computerized cognitive rehabilitation. Int J Med Inform. 2018 Jul;115:64-72. doi: 10.1016/j.ijmedinf.2018.04.005. Epub 2018 Apr 21. PMID 29779721
- [Background] Alloni A, Sinforiani E, Zucchella C, Sandrini G, Bernini S, Cattani B, Pardell DT, Quaglini S, Pistarini C. Computer-based cognitive rehabilitation: the CoRe system. Disabil Rehabil. 2017 Feb;39(4):407-417. doi: 10.3109/09638288.2015.1096969. Epub 2015 Oct 27. PMID 26505323
- [Derived] Bernini S, Panzarasa S, Barbieri M, Sinforiani E, Quaglini S, Tassorelli C, Bottiroli S. A double-blind randomized controlled trial of the efficacy of cognitive training delivered using two different methods in mild cognitive impairment in Parkinson's disease: preliminary report of benefits associated with the use of a computerized tool. Aging Clin Exp Res. 2021 Jun;33(6):1567-1575. doi: 10.1007/s40520-020-01665-2. Epub 2020 Sep 8. PMID 32895890